CLINICAL TRIAL: NCT03706144
Title: Evaluating Feasibility and Effectiveness of Computerized Mathematic Training - A Randomized Controlled Trial
Brief Title: Evaluating Feasibility and Effectiveness of Computerized Mathematic Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Julia Jaekel, Associate Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UTK IRB-18-04338-XM
Record Dates: First submitted 2018-10-05; First posted 2018-10-15 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Math Teachers (Grades 2-8); Math Students (Grades 2-8)

STUDY DESIGN:
Intervention Model Description: This is a randomized trial with two arms. Teachers (and their respective classes of students) have been randomized into one of two groups:
  1. Participating in the adaptive, online Prodigy Math Training
  2. treatment as usual (TAU) - classic math instruction in school
Who Masked: Outcomes Assessor
Masking Description: The primary outcomes are standardized, computerized assessments.
  Please note that the primary outcome is on the individual student level, while the randomization and participant number below is per teacher.
  Each teacher participates with 1-4 classes of on average 25 students
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prodigy Intervention Group (Experimental): Teachers will use the Prodigy Math Training with their students in school for at least 20 minutes per day, 3 days per week, from August to December 2018.
  Interventions: Other: Prodigy Math Training
- Control Group (No Intervention): Instruction as usual = TAU

INTERVENTIONS:
Other: Prodigy Math Training — https://www.prodigygame.com/
  Arms: Prodigy Intervention Group

SUMMARY:
This is a randomized controlled trial that is carried out in collaboration with Knox County Schools, using an adaptive, open-access, online math training programs as intervention and student growth in math attainment as the primary outcome over one school year.

DETAILED DESCRIPTION:
Computational fluency and understanding of mathematical concepts are essential for students' math achievement. Attainment of math learning goals in childhood uniquely predicts life-course success and wellbeing.Thus, investing in childhood math proficiency is critically important to prepare students for solving problems and succeeding in life. In schools, math teachers are faced with increasingly complex demands but instruction time is limited. Students who are struggling may need extensive individualized practice to succeed. To that end, novel computerized training methods are used in today's schools to help students obtain crucial abilities. According to the National Association for the Education of Young Children (NAEYC), most schools have adopted digital tools in the classroom, and they are increasingly interested in providing students access to new educational resources. Such specialized programs may have the potential to enhance children's academic growth trajectories, but they are not sufficiently evaluated. Moreover, teachers may not be prepared to select and use adequate digital tools.

There are numerous online learning programs that elicit different levels of motivation in students while adhering to Common Core State Standards. Some of them are expensive for schools whereas others are free, which makes them especially attractive for socioeconomically disadvantaged areas. One of the newer, but highly used programs is Prodigy, an adaptive open-access online math training game that continuously adapts to students' progress. Prodigy is different than most other programs because of its play-based, virtual reality environment that students explore with an avatar while solving math questions. As a result, students may be highly motivated and elect to spend more time on Prodigy than on other learning programs. Prodigy is currently being used by around 26 million students and teachers in the United States and Canada (https://www.prodigygame.com/), 150 school districts in the US have implemented Prodigy as part of their math curriculum, and many districts are expected to change from other programs to Prodigy, but the program has not been evaluated so far.

The investigators' aim is to evaluate the use and effectiveness of the adaptive Prodigy math training program via a randomized controlled trial (RCT) in the Knox County Schools (KCS) district.

ELIGIBILITY:
Inclusion Criteria:

* Elementary and middle school math teachers
* Students grades 2-8

Exclusion Criteria:

n/a

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Change in mathematic achievement | 8 months
  Change in mathematic achievement trajectories assessed with standardized Aimsweb Concepts and Applications scales test scores at three defined time points over 8 months: baseline (pre-test) assessment is in September, post-test and follow-up assessments take place in early January and late April 2019. An increase in scores indicates better outcomes (i.e., positive change) over time.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Jaekel, PhD, Principal Investigator — University of Tennessee Knoxville
Locations (1):
- University of Tennessee Knoxville, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No